CLINICAL TRIAL: NCT02392260
Title: Non-invasive Screening of the Status of the Vascular System: Feasibility Test
Acronym: NISTAS1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Valentina Favalli, Biomedical Engeneer, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 20140008054
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: To Evaluate the Validity of the Measure Method, we Will Compare Vasculight v1.0 PWV Measures With Those Obtained From E-tracking (Echocardiographic Method).

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vasculight prototype zero level (Experimental)
  Interventions: Device: Vasculight

INTERVENTIONS:
Device: Vasculight — Comparative measre of Pulse Wave velocity with both Vasculight prototype and Echocardiographic machine.

SUMMARY:
This project is part of the EU funded project NISTAS. NISTAS aims at the development of a new medical device for non-contact, non-invasive screening of the health status of the vascular system of adult subjects. The instrument, called VascuLight, is intended to be deployed at out-patient points-of-care and hospitals, and it provides output parameters related to the PWV as measured at local and/or at regional level.

NISTAS brings together four European SMEs in four different, but complementary, technology areas (JULIGHT, ECLEXYS, EPI-LIGHT, OIP) and links them with five RTD Performers (UNIPV, OSM, CORK UNIVERSITY, Saphyrion, Eudax srl ) to develop new knowledge and a new medical device which will have significant commercial benefits for all of the SME partners.

VascuLight responds to an unmet need in the medical diagnosis practice: the request for a fast and sustainable method for the screening of the health of the vascular system in large series, capable of providing a reliable indicator of the cardiovascular risk of the screened subjects.

The VascuLight idea is founded on a paradigm shift: bringing and adapting to the biomedical field measurement techniques that are to date confined to the industrial environment. NISTAS will develop new non-contact distance/displacement/vibration sensors based on a variant of the well-known and reliable laser triangulation technique.

JUL and UNIPV have carried out proof-of-concept, in-vivo tests of the VascuLight approach to demonstrate that the concept is realistic and attainable. Results have been obtained using Laser Doppler Vibrometry (LDV), a displacement-measuring technique based on the principle of light interference, and an area where both JUL and UNIPV have made important contributions. In the tests it was possible to use TWO small LDV optical heads to simultaneously measure the pulse wave in two points on the carotid spaced by 2.5 cm, allowing for the calculation of the time-delay between the pulse waves, and thus providing a direct local measurement of the PWV.

The aim of the study is to test the implemented contactless optical technique for the measurement of the PWV and the arterial stiffness at the carotid artery level.

To evaluate the validity of the measure method, the investigators will compare Vasculight v1.0 PWV measures with those obtained from e-tracking (echocardiographic method) . The main idea is to compare the distribution of measures (comparable mean and standard deviation) in the same mixed adult population, using the two different methods.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65

Exclusion Criteria:

1. Systolic BP >160 mmHg or diastolic BP >100 mmHg
2. Treated hypertension
3. Diagnosis of type 1 or type 2 diabetes mellitus
4. Treated hypercholesterolaemia
5. Past or current, symptomatic or proven, coronary artery disease
6. Clinical cerebrovascular disease
7. Carotid arterial stenosis
8. Severe peripheral vascular disease
9. Hypertrophic or dilated cardiomyopathy
10. Congestive heart failure
11. Heart valve disease
12. Previous cardiac surgery
13. Congenital heart disease
14. Other systemic diseases such as cancers, endocrine diseases and autoimmune diseases
15. Any regular drug treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Pulse Wave velocity | 1 month
  Bland Altmann test and ROC analysis will be used to compare the 2 methods